CLINICAL TRIAL: NCT07037043
Title: Hydrocortisone Plus Fludrocortisone in High-risk Patients Undergoing for Cardiac Surgery
Acronym: VASOCORT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2024_843_0047
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Inflammation in Cardiac Surgery
Keywords: Control of inflammation in cardiac surgery
MeSH Terms: interventions — Hydrocortisone; Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrocortisone plus fludrocortisone (Experimental): * Hydrocortisone 200 mg/day for 5 days or until ICU discharge, starting at the initiation of cardiopulmonary bypass (CPB), administered intravenously via syringe pump in a double-blind manner
  * Fludrocortisone 50 µg/day in the morning for 5 days or until ICU discharge, administered orally or via nasogastric tube (if the patient is sedated), diluted in a glass of water, in a double-blind manner
  Interventions: Drug: hydrocortisone plus fludrocortisone
- placebo of hydrocortisone plus fludrocortisone (Placebo Comparator): * Placebo for hydrocortisone (0.9% NaCl) administered following the same protocol as fludrocortisone in the intervention group
  * Placebo for fludrocortisone (capsule containing microcrystalline cellulose diluted in a glass of water) administered following the same protocol as fludrocortisone in the intervention group
  Interventions: Drug: placebo of hydrocortisone plus fludrocortisone

INTERVENTIONS:
Drug: hydrocortisone plus fludrocortisone — * Hydrocortisone 200 mg/day for 5 days or until ICU discharge, starting at the initiation of cardiopulmonary bypass (CPB), administered intravenously via syringe pump in a double-blind manner
  * Fludrocortisone 50 µg/day in the morning for 5 days or until ICU discharge, administered orally or via nasogastric tube (if the patient is sedated), diluted in a glass of water, in a double-blind manner
  Arms: hydrocortisone plus fludrocortisone
Drug: placebo of hydrocortisone plus fludrocortisone — * Placebo for hydrocortisone (0.9% NaCl) administered following the same protocol as fludrocortisone in the intervention group
  * Placebo for fludrocortisone (capsule containing microcrystalline cellulose diluted in a glass of water) administered following the same protocol as fludrocortisone in the intervention group
  Arms: placebo of hydrocortisone plus fludrocortisone

SUMMARY:
Cardiac surgery is a high-risk surgery and is associated with a rate of postoperative adverse outcomes. Like many others major surgery, cardiac surgery procedures induce a proinflammatory phase usually counterbalanced with an immunosuppressive phase so the immune response remained balanced.

In some cases, the immune response might be dysregulated with a more pronounced pro inflammatory state that compromises organ perfusion and with the occurrence of organ failure. From a mechanistic approach, the relationship between organ failure is complex and multifactorial with a high level of proinflammatory cytokines, a decrease in microcirculation, an endothelial dysfunction and an activation of coagulation and over. The clinical expression is an increase in vasopressor exposure and dose, an increase in mortality and in adverse outcomes with a predominance of acute kidney injury.

Various therapies have been assessed to manage cardiac surgery related sepsis including glucocorticoid therapy. Briefly, two major randomized trials assessed glucocorticoid therapy solely in scheduled cardiac surgery with cardiopulmonary bypass. No clinical benefit was demonstrated in term of reduction in postoperative mortality or adverse outcomes. Since, data support that the selection of patients at risk is crucial to demonstrate such a strategy. Indeed, data support that surprisingly some patients will have a very light immune response reflected by a low pro inflammatory cytokine.

The hypothesis is that the combination glucocorticoid and fludrocortisone could decrease adverse outcomes in selected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patient at intermediate/high risk (EuroSCORE II > 4%).
* Patient admitted for scheduled cardiac surgery:

  * Coronary artery bypass grafting (CABG).
  * Aortic valve replacement.
  * Mitral valve repair or replacement.
  * Surgery of the aortic root (aortic tube, Bentall procedure, Tirone David procedure, or other).
  * Combined surgery.
* Patient undergoing cardiopulmonary bypass (CPB).
* Informed consent signed by the patient.

Exclusion Criteria:

* Endocarditis
* Off-pump heart surgery
* Heart transplantation or long-term ventricular assist device (VAD)
* Emergency surgery: aortic dissection, emergency coronary artery bypass grafting (CABG)
* Failure to wean from CPB requiring short-term mechanical support (intra-aortic balloon pump, ECMO)
* Hypothermic surgery
* History of cardiac surgery
* Patient on long-term corticosteroid therapy
* Autoimmune disease or chronic inflammatory condition
* End-stage renal disease on long-term dialysis
* Contraindications to the administration of hydrocortisone and/or fludrocortisone according to the summary of product characteristics (SmPC)
* Pregnant or breastfeeding woman
* Patient under legal protection (guardianship, curators, or judicial safeguard).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Variation of acute kidney injury occurence between both groups | up to 7 days
Variation of postoperative pulmonary complication occurrence between both groups | up to 7 days
Variation of number of norepinephrine requirement between both groups | up to 7 days

SECONDARY OUTCOMES:
variation of postoperative atrial fibrillation occurence between both groups | up to 7 days
  Postoperative atrial fibrillation: defined as a new-onset arrhythmia within 7 days after surgery, documented by an electrocardiogram showing absence of P waves and narrow, irregular QRS complexes
variation of myocardial infarction occurence between both groups | up to 7 days
  Myocardial infarction: defined according to the Fourth Universal Definition
variation of stroke occurence between both groups | up to 7 days
  Stroke: defined as the sudden onset of a neurological deficit confirmed by brain imaging
Variation of total amount of norepinephrine between both groups | up to 7 days
  The total amount of norepinephrine will be expressed in milligrams and will correspond to the cumulative dose administered from ICU admission until the 7th postoperative day.
variation of occurrence of glucocorticoid side effect between both groups | up to 7 days
  glucocorticoid side effects are hyperglycemia, hypernatremia and infections
Variation of 28-day mortality between both groups | at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No